CLINICAL TRIAL: NCT01093131
Title: Oral Hydration and Alkalinization is Non-Inferior to Intravenous Therapy for Prevention of Contrast Induced Nephropathy in Patients With Chronic Kidney Disease.
Brief Title: Oral Versus Intravenous Hydration to Prevent Contrast Induced Nephropathy
Acronym: HYDRATE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: The Western Pennsylvania Hospital (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 04-11-097-DT / WPCI 2009-28
Record Dates: First submitted 2010-02-25; First posted 2010-03-25 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2016-11

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast induced nephropathy; Percutaneous transluminal coronary angioplasty; chronic kidney disease; Prevention; Equivalence
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intravenous Hydration (Active Comparator): Pretreatment with a 3 mL/kg bolus of intravenous normal saline solution (154 mEq/L) over 1 hour, immediately prior to contrast exposure followed by intravenous infusion of 1ml/kg per for 6 hours after the procedure.
  Interventions: Other: Intravenous Hydration
- Intravenous hydration and sodium bicarbonate (Active Comparator): Pretreatment with a 3 mL/kg bolus of intravenous sodium bicarbonate solution (154 mEq/L) over 1 hour, immediately prior to contrast exposure followed by intravenous infusion of 1 mL/kg for 6 hours after the procedure.
  Interventions: Other: Intravenous Hydration; Drug: Intravenous sodium bicarbonate
- Oral hydration (Active Comparator): Oral hydration with 500 mL of water to be started 4 hours prior to contrast exposure and stopped 2 hours prior to procedure followed by oral hydration with 600 mL of water post procedure
  Interventions: Other: Oral hydration
- Oral hydration and oral sodium bicarbonate (Active Comparator): Oral hydration with 500 mL of water to be started 4 hours prior to procedure and stopped 2 hours prior to contrast exposure, with the addition of 3.9 grams (46.4 mEq) of oral sodium bicarbonate to be given 20 minutes prior to contrast exposure followed by 1.95 grams (30.4 mEq) of oral sodium bicarbonate 2 hours and 4 hours after the initial dose
  Interventions: Other: Oral hydration; Drug: Oral sodium bicarbonate

INTERVENTIONS:
Other: Oral hydration — Oral hydration with 500 mL of water to be started 4 hours prior to contrast exposure and stopped 2 hours prior to procedure followed by oral hydration with 600 mL of water post procedure
  Arms: Oral hydration; Oral hydration and oral sodium bicarbonate
Drug: Oral sodium bicarbonate — Oral hydration with 500 mL of water to be started 4 hours prior to procedure and stopped 2 hours prior to contrast exposure, with the addition of 3.9 grams (46.4 mEq) of oral sodium bicarbonate to be given 20 minutes prior to contrast exposure followed by 1.95 grams (30.4 mEq) of oral sodium bicarbonate 2 hours and 4 hours after the initial dose
  Arms: Oral hydration and oral sodium bicarbonate
Other: Intravenous Hydration — Pretreatment with a 3 mL/kg bolus of intravenous normal saline solution (154 mEq/L) over 1 hour, immediately prior to contrast exposure followed by intravenous infusion of 1ml/kg per for 6 hours after the procedure.
  Arms: Intravenous Hydration; Intravenous hydration and sodium bicarbonate
Drug: Intravenous sodium bicarbonate — Pretreatment with a 3 mL/kg bolus of intravenous sodium bicarbonate solution (154 mEq/L) over 1 hour, immediately prior to contrast exposure followed by intravenous infusion of 1 mL/kg for 6 hours after the procedure.
  Arms: Intravenous hydration and sodium bicarbonate

SUMMARY:
The increased risk for contrast-induced nephropathy (CIN) in patients with chronic kidney disease (CKD) undergoing coronary angiography (CAG) has been established. Current and historical data on CIN prevention strategies have shown wide variation with respect to the optimal type, route and timing of these therapies. We investigate the role for oral hydration and/or oral sodium bicarbonate administration compared to intravenous hydration and/or sodium bicarbonate in patients with CKD undergoing CAG.

DETAILED DESCRIPTION:
This is a single center study randomizing patients with CKD undergoing CAG into 4 groups: 1) Intravenous normal saline, 2) Intravenous normal saline and intravenous bicarbonate, 3) oral hydration, and 4) oral hydration and oral bicarbonate. The primary endpoint was the occurrence of contrast-medium-induced nephropathy defined as greater than 25% increase in serum creatinine from baseline or an absolute increase of 0.5 mg/dL from baseline at 72 hours following exposure to radiocontrast. Secondary endpoints include the length of hospitalization and in-house mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Stable serum creatinine levels of at least 1.1 mg/dL or estimated creatinine clearance less than 60 mL/min
2. Scheduled for diagnostic, elective cardiac angiography

Exclusion Criteria:

1. Serum creatinine levels >8.0 mg/dL
2. Change in serum creatinine levels of at least 0.5 mg/dL during the previous 24 hours
3. Preexisting dialysis
4. Multiple myeloma or other myeloproliferative disease
5. Current CHF or recent history of flash pulmonary edema
6. Current myocardial infarction
7. Symptomatic hypokalemia
8. Uncontrolled hypertension (treated systolic blood pressure >200 mmHg or diastolic blood pressure >100mmHg)
9. Exposure to radiocontrast within 7 days the study
10. Emergency Catheterization
11. Allergy to radiographic contrast
12. Pregnancy
13. Administration of dopamine, mannitol, fenoldapam, or N-acetylcysteine during the time of the study
14. Severe COPD
15. Serum Bicarb > 28
16. Sodium <133

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-02; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Contrast Induced Nephropathy | 72 hours
  Defined as greater than 25% increase in serum creatinine from baseline or an absolute increase of 0.5 mg/dL from baseline at 72 hours.

SECONDARY OUTCOMES:
Length of Hospital Stay | 72 hours
  Defined as number of days in the hospital.
In-Hospital Mortality | 72 hours
  Any cause of mortality
Aspiration | 72 hours
  Defined as oxygen saturation less than 92% by pulse oximetry.
Hypotension | 72 hours
  Defined as a systolic blood pressure less than 100 mmHg by conventional measuring methods.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Cho, MD MHSA, Study Director — The Western Pennsylvania Hospital
Locations (1):
- The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania, United States